CLINICAL TRIAL: NCT04206215
Title: Noninvasive Brain Stimulation for Treating Carpal Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Highland Instruments, Inc. (Industry)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019P002804
Record Dates: First submitted 2019-12-02; First posted 2019-12-20 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain; Carpal Tunnel Syndrome
Keywords: transcranial Direct Current Stimulation; Transcranial Ultrasound; Noninvasive brain stimulation
MeSH Terms: conditions — Chronic Pain; Carpal Tunnel Syndrome | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active tDCS + Active TUS (Experimental): Subjects in the experimental group will undergo 20 minutes of active transcranial direct current stimulation (tDCS) and active transcranial ultrasound (TUS).
  Interventions: Device: transcranial Direct Current Stimulation (tDCS); Device: Transcranial Ultrasound (TUS)
- Sham tDCS + Sham TUS (Sham Comparator): Subjects in the sham group will undergo 20 minutes of sham transcranial direct current stimulation (tDCS) and sham transcranial ultrasound (TUS).
  Interventions: Device: transcranial Direct Current Stimulation (tDCS); Device: Transcranial Ultrasound (TUS)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2mA. In the sham group, the tDCS device will not be active for the full 20 minutes.
Device: Transcranial Ultrasound (TUS) — Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.

SUMMARY:
The purpose of this study is to assess the effects of tDCS in combination with TUS for the treatment of pain in subjects with Carpal Tunnel Syndrome. The investigators hypothesize that there will be a decrease in pain levels with active stimulation, when compared to sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent to participate in the study
2. Subjects between 18 to 80 years old
3. Having symptomatic CTS spreading within or beyond the median nerve distribution (demonstrating 'extra-median spread'), involving at least 1 wrist, with chronic pain as defined by International Association for the Study of Pain (existing pain for at least 6 months and having pain on at least half the days in the past 6 months with an average of at least a 3 on a 0-10 VAS scale).
4. Pain resistant to first line therapies of chronic pain (pain still present at lower levels most of the time following therapy)
5. Must have the ability to feel pain as self-reported.

Exclusion Criteria:

1. Subject is pregnant
2. Contraindications to tDCS+TUS:

   1. intracranial metal implant
   2. implanted brain medical devices
3. History of alcohol or drug abuse within the past 6 months as self-reported
4. Use of carbamazepine within the past 6 months as self-reported
5. Suffering from major depression (with a PHQ-9 score of ≥20)
6. History of neurological disorders involving stroke, brain tumors, or epilepsy with residual neurological symptoms as self-reported (note patients will also be evaluated via EEG at baseline about 1 week prior to stimulation and any patient showing abnormal EEG activity will be removed))
7. History of unexplained fainting spells as self-reported
8. History of head injury resulting in more than a momentary loss of consciousness as self-reported and with current neurological deficits
9. History of intracranial neurosurgery as self-reported

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2025-10-06 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS) | 9 weeks
  Changes in the Visual Analogue Scale (VAS) for pain will be measured in order to determine whether anodal transcranial direct current stimulation in conjunction with transcranial ultrasound is effective in reducing pain in subjects with Carpal Tunnel Syndrome.
  The VAS scale goes from 0 up to 10, where 0 means no pain at all and 10 means the worst imaginable pain.

SECONDARY OUTCOMES:
Verbal Rating Scale (VRS) | Measured for approximately for a total 9 weeks
  Changes in the Verbal Rating Scale (VRS) for pain will be measured in order to determine whether anodal transcranial direct current stimulation in conjunction with transcranial ultrasound is effective in reducing pain in subjects with Carpal Tunnel Syndrome. The VRS minimum value is no pain and the maximum value is severe pain. Being severe pain the worst outcome.
Visual Analog Mood Scale (VAMS) | Measured for approximately for a total 9 weeks
  The investigators will measure safety of tDCS and TUS by measuring changes in the Visual Analog Mood Scale.
  This scale will range from zero (low or worst mood) to 10 on anxiety, depression, sleepiness and stress.
Montreal Cognitive Assessment (MOCA) | Measured for approximately for a total 9 weeks
  The investigators will monitor the safety of tDCS and TUS in subjects by measuring any changes in cognition, attention, and focus with the MOCA. MOCA scores range between 0 and 30, a score of 26 and higher generally considered normal.
tDCS Side Effects Questionnaire | Measured for approximately for a total 9 weeks
  At each session, subjects will complete a questionnaire to evaluate potential adverse effects of stimulation (headache, neck pain, mood alterations, and seizures) on a 4-point scale, where 1 is absent and 4 is severe. The scale will also be administered at the follow-ups.
Patient Health Questionnaire (PHQ-9) | Measured for approximately for a total 9 weeks
  The investigators will measure safety of tDCS and TUS by measuring changes of mood through the PHQ-9. The scoring goes from 0 to 27, where 0 is no depression and 27 is severe depression.
Multidimensional Pain Inventory (MPI) | Measured for approximately for a total 9 weeks
  The investigators will monitor the impact of pain with the MPI of tDCS and TUS. It consist in 3 sections (Pain Impact , responses by significant others, activities and each item is rated on a 7-point scale (0-6), where higher scores represent severe symptoms .
Neuropathic Pain Symptom Inventory (NPSI) | Measured for approximately for a total 9 weeks
  The investigators will monitor the changes of neuropathic pain in subjects going through the study before and after tDCS and TUS. It include 12 items in total, this tool evaluates mean pain intensity in the last 24 hours in a numeric scale from zero (no pain) to 10 (worst imaginable pain). Total pain intensity score may be calculated by the sum of 10 descriptors
Temporal Summation (TS) | Measured for approximately for a total 9 weeks
  The investigators will monitor the changes of temporal summation in the study before and after tDCS and TUS. This will be assessed by Von Frey filaments. This is assessed by having the participant rate their pain after a single stimulus (6.65, 300 g) applied for 0.5 s and then again after a series of 10 (6.65, 300 g) stimuli are applied at 1-s intervals.
Conditioned pain modulation (CPM) | Measured for approximately for a total 9 weeks
  Changes in the conditioned pain modulation will be measured in order to determine whether anodal transcranial direct current stimulation in conjunction with transcranial ultrasound is effective in changing the conditioned pain modulation system in subjects with Carpal Tunnel Syndrome. This will be assessed by applying pressure with an algometer.
Vibration Detection Threshold (VDT) | Measured for approximately for a total 9 weeks
  Changes in the vibration detection threshold will be measured , this is performed with a Rydel-Seiffer tuning fork (64 Hz, 8/8 scale) placed on the skin surface and is determined by asking the participant to tell the examiner when the vibration is no longer felt.
Michigan Hand Outcomes Questionnaire (MHQ) | Measured for approximately for a total 9 weeks
  This a hand-specific outcomes instrument that measures outcomes of patients with conditions of, or injury to, the hand or wrist. The MHQ contains six distinct scales: overall hand function, activities of daily living , pain, work performance, aesthetics, and patient satisfaction with hand function. They are scored from 0 - 100 in which 100 is the best possible ability
Boston Carpal Tunnel Questionnaire | Measured for approximately for a total 9 weeks
  This is an instrument specifically designed for Carpal Tunnel Syndrome (CTS) and validated for CTS therapy assessments (consisting of the Functional Status Scale and Symptom Severity Scale scores. The symptom severity scale has 11 questions scored from 1 point (mildest) to 5 points (most severe).
The Medical Outcomes Study 36-Item Short Form (SF-36) | Measured for approximately for a total 9 weeks
  This a generic health status instrument that measures 8-health related concepts using 36 questions and provides a profile of functional health and well-being scores. It also provides a psychometrical index of physical and mental health. Each scale is transformed into a 0-100 scale. The lower the score the more disability. The higher the score the less disability
Electroencephalography (EEG) | Measured for approximately for a total 3 weeks
  Investigators will measure electroencephalogram activity to monitor safety. Baseline recordings will be reviewed to ensure that there are no potential electroencephalographic safety criteria prior to stimulation. This qualitative analysis will focus on pathological EEG activity such as epileptiform discharges or persistent focal slowing.
Strength (grip and pinch) | Measured for approximately for a total 9 weeks
  Strength will be assessed using a grip dynamometer and a pinch dynamometer
Range of Motion (ROM) | Measured for approximately for a total 9 weeks
  The investigators will assess active and passive ROM in the elbow, forearm, wrist, thumb, digits
Thumb Reaching Test | Measured for approximately for a total 9 weeks
  Subject will be asked to reach the base of the little finger with their thumb. The task will be repeated up to 10 times. Primary data will be taken from inertial sensors placed on the thumb and little finger.
Reach to Pinch | Measured for approximately for a total 9 weeks
  Subject will be asked to perform a reach to pinch task . The task will be repeated up to 10 times. Primary data will be taken from camera and accelerometers/gyroscopes placed on the thumb and index finger.
Wrist Flexion-Extension: | Measured for approximately for a total 9 weeks
  Subject will be asked to flex-extend their wrist up to 10 times. Primary data will be taken from an accelerometer/gyroscope placed on the wrist and the camera.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD PhD MPH, Principal Investigator — Spaulding Rehabilitation Network
Locations (1):
- Spaulding Rehabilitation Network Research Institute, Charlestown, Massachusetts, United States